CLINICAL TRIAL: NCT00675753
Title: Genetic Variations in Three Interacting Single Nucleotide Polymorphisms and the Risk of Preterm Birth in Black Families
Brief Title: Three Interacting Single Nucleotide Polymorphisms (SNPs) and the Risk of Preterm Birth in Black Families
Status: Terminated | Type: Observational
Why Stopped: Study site did not have sufficient subjects for the case group
Sponsor: University of Miami (Other)
Collaborators: Pediatrix (Other)
Responsible Party: Principal Investigator, Victoria Mitrani, Professor, University of Miami
Other Study IDs: 20070609
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Premature Birth
Keywords: Genes; Ethnology; Cytokines; prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood spot specimens were collected from the mother and her infant.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preterm group: Preterm (36 6/7 weeks gestation or earlier) mothers and their newborns.
  Interventions: Genetic: Blood spot specimens will be drawn
- Term group: Term (> 37 weeks gestation) mothers and their newborns.
  Interventions: Genetic: Blood spot specimens will be drawn

INTERVENTIONS:
Genetic: Blood spot specimens will be drawn — Blood spot specimens will be drawn from mother-baby dyads in the control and experimental groups and sent for genotyping
  Other Names: High risk genetic combinations; Low risk genetic combinations

SUMMARY:
A multilocus interaction of three pro-inflammatory cytokine single nucleotide polymorphisms (SNPs), -3448 Tumor Necrosis Factor-α, -7227 Interleukin 6, and 33314 Interleukin 6R was reported by Menon and associates in 2006. The researchers reported that they were able to predict spontaneous preterm birth in 65.2% of a population restricted to European-American mothers. Expansion of this research is needed to determine if the results are also applicable in Black populations.

Statement of Purpose The purpose of this research is to determine if the multi-locus genetic interaction of tumor necrosis factor-α (-3448), interleukin 6 (-7227), and interleukin 6R (33314), as described by Menon et al. (2006), is associated with preterm birth in Black mother-infant dyads.

Research Aims and Hypotheses:

Primary Aim 1.0: To determine if carriage of one of the high risk genetic patterns, as identified by Menon et al. (2006), is present in 65% of Black mothers with preterm births and 35% of Black mothers with term births.

Hypothesis 1.0: There is no statistically significant difference in the occurrence of one of the eight high risk genetic patterns, as identified by Menon et al. (2006), in a population of Black mothers with preterm births (case) and Black mothers with term births (controls).

Primary Aim 2.0: To determine if carriage of one of the high risk genetic patterns, as identified by Menon et al. (2006), is present in 65% of Black preterm newborns and 35% of Black term newborns.

Hypothesis 2.0: There is no statistically significant difference in the occurrence of one of the eight high risk genetic patterns, as identified by Menon et al. (2006), in a population of Black preterm newborns (case) and Black term newborns (controls).

DETAILED DESCRIPTION:
Research Design and Methods

Study Design A gene association study, using a case-control design, will be utilized. Each case and each control will include the genetic mother and her newborn infant.

Setting A multicenter (n=2) study is proposed. St. Mary's Medical Center in West Palm Beach, Florida and Broward General Medical Center in Ft. Lauderdale, Florida are the two research centers.

Sample:

It is estimated that a sample of 166 mother-infant dyads (332 individuals) will be needed to test the study hypotheses. The sample size has been adjusted to allow for a 10% drop out rate. The control group will include 110 term mothers and 110 term infants. The case group will include 56 preterm mothers and 56 preterm infants.

It is expected that each site will be able to enroll 83 family dyads in less than two years. A reasonable effort will be made to enroll eligible family dyads. Enrollment of less than 50% of eligible subjects will lead to a site review to remedy the problem or result in possible site closure. Enrollment for each site will be a minimal of 66 family dyads and a maximum of 100 family dyads.

ELIGIBILITY:
Inclusion Criteria:

* Mother and Father, if named on the birth certificate application, are English speaking.
* If mother and Father are married, husband is the man identified as the father on the birth certificate application.
* Documentation of Informed Consent for Mother and newborn. Father named on the birth certificate application must consent for newborn to participate.
* Mother's age (and Father if named on the birth certificate application) is 18 years of age or older.
* Infant is a singleton, inborn newborn.
* Newborn gestational age assessment documented in the health record between 23 weeks 0/7 days and 36 weeks 6/7 days.
* Newborn gestational age assessment documented in the health record > 37 weeks and 0/7 days.
* Mother identifies herself as Black or African American on the birth certificate application.

Exclusion Criteria:

* Mother (or Father identified on the birth certificate application) refuses to sign informed consent.
* Mother (or Father identified on the birth certificate application) does not speak English.
* Father, identified on the birth certificate application, objects to infant's participation.
* Husband is not the father named on the birth certificate application.
* Mother (or Father, if named on the birth certificate application) is less than 18 years of age.
* Mother fails to identify her ethnic group as Black or African American on the birth certificate application.
* Mother is cognitively impaired as a result of receiving narcotic analgesia within four hours of the time the research is explained, consent explained, or the interview is conducted.
* Mother is documented to be cognitively impaired by her physician in the medical record.
* Father appears to be cognitively impaired at the time the research is explained, consent explained, or the interview is conducted.
* Mother or infant has a history of blood transfusion in the last six months.
* Mother had assisted reproduction.
* Maternal surgical procedures during pregnancy, to include cerclage.
* Mother has uterine abnormalities.
* History of trauma prior to the onset of labor.
* Multiple gestation.
* Infant has major anomalies (cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia or other major gastrointestinal anomalies, major neurological injury or anomaly, or multiple congenital anomalies).
* Mother has major anomalies (cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia or other major gastrointestinal anomalies, major neurological injury or anomaly, or multiple congenital anomalies).
* Infant has documented chromosomal anomalies.
* Mother has documented chromosomal anomalies.

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study populations were preterm mothers and their infants, born prior to 37 weeks gestation, and term mothers and their infants.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine if carriage of one of the high risk genetic patterns, as identified by Menon et al. (2006), is present in 65% of Black mothers and their infants with preterm births and 35% of Black mothers and their infants with term births. | 2 years

SECONDARY OUTCOMES:
To determine the frequency of low risk genetic patterns, as identified by Menon et al. (2006), in Black mothers and their infants with preterm births and Black mothers and their infants with term births. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gail McCain, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Broward Medical Center, Fort Lauderdale, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida

REFERENCES:
- [Background] Menon R, Velez DR, Simhan H, Ryckman K, Jiang L, Thorsen P, Vogel I, Jacobsson B, Merialdi M, Williams SM, Fortunato SJ. Multilocus interactions at maternal tumor necrosis factor-alpha, tumor necrosis factor receptors, interleukin-6 and interleukin-6 receptor genes predict spontaneous preterm labor in European-American women. Am J Obstet Gynecol. 2006 Jun;194(6):1616-24. doi: 10.1016/j.ajog.2006.03.059. PMID 16731080